CLINICAL TRIAL: NCT00503048
Title: Markers of Atopy in Children With Presumed Early Exposure to Allergens, Unhygienic Conditions, and Infections
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Iwona Stelmach MD, PhD, Prof, Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Other Study IDs: RNN-268-03-KE
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Atopic Diseases
Keywords: atopy; atopic diseases; children; orphanages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: foster care children
- 2: reference children (living with families)

SUMMARY:
There are many studies regarding possible causes of increasing trend in frequency of allergic diseases in the last three decades. Main causes of this trend are: decrease of infectious diseases frequency, improvement in life level, changes in diet and lactic acid bacterias elimination from digestive tract. Primary Purpose of this study is to compare the prevalence of atopy and atopic diseases in two child populations: foster care and reference children and - to define risk and protective factors for the development of atopy.

DETAILED DESCRIPTION:
There are many studies regarding possible causes of increasing trend in frequency of allergic diseases in the last three decades. Main causes of this trend are: decrease of infectious diseases frequency, improvement in life level, changes in diet and lactic acid bacterias elimination from digestive tract. Less exposition to microbes can lead to the disturbance in optimal balance between Th1 and Th2 lymphocytes, prevalence of Th2 cytokines and excessively high production of IgE. Decreased exposure to microbes has resulted in the loss of main source of immune provocation, and a consequent increase in pathogenic immune responses and their associated diseases. Molecular interactions between immunocytes and microbes are mediated largely by Toll-like receptors (TLRs) on host cells and a diversity of ligands produced by viruses, bacteria and fungi.

Many studies confirm the protective role of some viral, bacterial or parasite infections against atopy development.

The studied group consisted of 500 children, living in all the ten community foster homes in Lodz. The reference group consisted of 500 children, living with their parents at home, recruited from primary care centres.

Primary Purpose of this study is to compare the prevalence of atopy and atopic diseases in two child populations: foster care and reference children and - to define risk and protective factors for the development of atopy.

Secondary Purpose is the genotyping and cytometric study - to define risk and protective factors for the development of atopy.

Primary outcome measures: skin prick test results with 18 allergens, peripheral blood eosinophil count, level of total and specific IgE in children with positive skin-test results were secondary and point, spirometry, medical history and physical examination.

Secondary outcome measures: included symptoms of asthma and other allergic diseases, lung function, parental allergy only for children from reference group, family history including life conditions in very early childhood, and markers of allergy such as total IgE serum concentration and eosinophil blood count, expression of TLR2, TLR4, TLR7, TLR9, examining the serum samples for specific antibodies to Toxocara sp, Toxoplasma gondi, Ascaris lumbricoides, DNA.

ELIGIBILITY:
Inclusion Criteria:

* must be able to make spirometry

Exclusion Criteria:

* pregnancy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children.
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2003-12; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Smejda, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz Lodz, Poland, Lodz, Poland

REFERENCES:
- [Result] Stelmach I, Smejda K, Kaczmarek J, Stelmach W, Kuna P. [Prevalence of atopy and atopic diseases in children living in an orphanage in Lodz area--pilot study]. Pol Merkur Lekarski. 2006 May;20(119):531-4. Polish. PMID 16875155
- [Result] Stelmach I, Smejda K, Jerzynska J, Stelmach W, Majak P, Stelmach P, Kuna P. Decreased markers of atopy in children with presumed early exposure to allergens, unhygienic conditions, and infections. Ann Allergy Asthma Immunol. 2007 Aug;99(2):170-7. doi: 10.1016/S1081-1206(10)60641-2. PMID 17718105
- See also: Article - Ann Allergy Asthma Immunol. 2007 Aug;99(2):170-7. — http://www.ncbi.nlm.nih.gov/pubmed/17718105?ordinalpos=1&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum
- See also: Article - Pol Merkur Lekarski. 2006 May;20(119):531-4. — http://www.ncbi.nlm.nih.gov/pubmed/16875155?ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum